CLINICAL TRIAL: NCT05698082
Title: Monkeypox and Cancer: a Pan-cancer Based Multi-omics Analysis and Single Cell Sequencing Analysis-Experimental Studies
Brief Title: FOS Immunohistochemical Staining of Colorectal Cancer and Its Adjacent Tissues
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: xiaoliang Huang (Other)
Responsible Party: Sponsor-Investigator, xiaoliang Huang, clinical Professor, Cancer Hospital of Guangxi Medical University
Organization: Cancer Hospital of Guangxi Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: KY-2020-305
Record Dates: First submitted 2023-01-16; First posted 2023-01-26 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Colorectal Cancer; Monkey Pox
Keywords: Differential expression of gene; Immunohistochemical staining; Tumor microenvironment
MeSH Terms: conditions — Colorectal Neoplasms; Mpox, Monkeypox

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Test group-stained by FOS antibody (Experimental): Sixty colorectal cancer tissue sections were included. The tissue was cut to 5 μm thick and placed on a glass slide for staining. Endogenous peroxidase activity was inhibited and blocked by deparaffin, rehydration, and treatment with 5% bovine serum albumin for 30 min at 37 ° C. The treated sections were incubated with anti-FOS (promab 30360) overnight at 4 ° C and washed three times with PBS. After that, it was required to incubate with secondary anti-peroxidation sunflower for 30 min at 37 ° C. After washing three times with PBS, the images were developed in diamine benzidine and micrographs were obtained under a light microscope.
  Interventions: Diagnostic Test: Immunohistochemical staining with anti-FOS

INTERVENTIONS:
Diagnostic Test: Immunohistochemical staining with anti-FOS — The tissue sections were incubated with anti-FOS (promab 30360) at 4ºC overnight and washed three times with PBS. After that, it is required that incubation with secondary anti-peroxidation sunflower at 37ºC for 30 minutes. After washing three times again with PBS, the sections were developed in diaminobenzidine and microscopic images were made by light microscopy.

SUMMARY:
Colorectal cancer tissue sections were obtained according to the inclusion criteria. The formalin was used to immersed all cancer specimens. And tissues were cut to 5 μm thickness and placed on glass slides before staining. Endogenous peroxidase activity was inhibited and blocked by de-paraffinizing, rehydrating, and using 5% bovine serum albumin at 37ºC for 30 min. The treated sections were incubated with anti-FOS (promab 30360) at 4ºC overnight and washed three times with PBS. After that, it is required that incubation with secondary anti-peroxidation sunflower at 37ºC for 30 minutes. After washing three times again with PBS, the sections were developed in diaminobenzidine and microscopic images were made by light microscopy.

ELIGIBILITY:
Inclusion Criteria:

* (a) patients with histologically confirmed CRC (b) patients who underwent resection of the primary tumor (c) patients at first visit who had not received treatment before blood testing.

Exclusion Criteria:

* (a) familial adenomatous polyposis or hereditary colon cancer (b) no signs of clinical infection, such as fever, on the day of blood collection; And (c) patients with multiple primary tumors during hospitalization.

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Original survival | Participants were followed up for 3 years, including outpatient follow-up and telephone follow-up.
  Time from the start of the study to death from any cause. For subjects who were lost to follow-up before death, the time of last follow-up was calculated as the time of death.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangxi Medical University Cancer Hospital, Nanning, Guangxi, China

IPD SHARING:
Plan to Share IPD: No